CLINICAL TRIAL: NCT06212648
Title: A Multi-center, Randomized, Double-blind, Parallel, Phase 2 Clinical Trial to Compare and Evaluate the Efficacy and Safety of SPC1001 and Monotherapy in Patients With Essential Hypertension
Brief Title: Evaluate the Efficacy and Safety of SPC1001 and Monotherapy in Patients With Essential Hypertension
Acronym: SP-CAP-002
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shin Poong Pharmaceutical Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SP-CAP-002
Record Dates: First submitted 2022-11-14; First posted 2024-01-19 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Hypertension; Essential Hypertension
Keywords: SP-CAP-002
MeSH Terms: conditions — Hypertension; Essential Hypertension | interventions — candesartan; Amlodipine

STUDY DESIGN:
Intervention Model Description: This clinical trial is a randomized, double-blind, parallel design, placebo and active drug comparison, and multicenter clinical trial to evaluate the safety and efficacy of investigational drugs after 8 weeks of administration.
Who Masked: Participant, Investigator
Masking Description: double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- SPC1001 High (Experimental): SPC1001 High (Candesartan/Amlodipine/Indapamide)
  Interventions: Drug: SPC1001 High; Drug: Placebo
- SPC1001 Mid1 (Experimental): SPC1001 Mid1 (Candesartan/Amlodipine/Indapamide)
  Interventions: Drug: SPC1001 Mid1; Drug: Placebo
- SPC1001 Mid2 (Experimental): SPC1001 Mid1 (Candesartan/Amlodipine/Indapamide)
  Interventions: Drug: SPC1001 Mid2; Drug: Placebo
- SPC1001 Low (Experimental): SPC1001 Low (Candesartan/Amlodipine/Indapamide)
  Interventions: Drug: SPC1001 Low; Drug: Placebo
- SPC3001 (Active Comparator): SPC3001 (Candesartan 8mg)
  Interventions: Drug: SPC3001; Drug: Placebo
- SPC4001 (Active Comparator): SPC4001 (Amlodipine 5mg)
  Interventions: Drug: SPC4001; Drug: Placebo
- SPC4002 (Active Comparator): SPC4002 (Amlodipine 10mg)
  Interventions: Drug: SPC4002; Drug: Placebo
- Placebo (Placebo Comparator): SPC1001(High, Mid1, Mid2, Low) placebo, SPC3001 placebo, SPC4001 placebo, SPC4002 placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SPC1001 High — Drugs for clinical trials are orally administered once a day after breakfast.
  After randomization, the drug for clinical trials is taken once a day (total of 4 tablets) for 8 weeks.
  Arms: SPC1001 High
Drug: SPC1001 Mid1 — Drugs for clinical trials are orally administered once a day after breakfast.
  After randomization, the drug for clinical trials is taken once a day (total of 4 tablets) for 8 weeks.
  Arms: SPC1001 Mid1
Drug: SPC1001 Mid2 — Drugs for clinical trials are orally administered once a day after breakfast.
  After randomization, the drug for clinical trials is taken once a day (total of 4 tablets) for 8 weeks.
  Arms: SPC1001 Mid2
Drug: SPC1001 Low — Drugs for clinical trials are orally administered once a day after breakfast.
  After randomization, the drug for clinical trials is taken once a day (total of 4 tablets) for 8 weeks.
  Arms: SPC1001 Low
Drug: SPC3001 — Drugs for clinical trials are orally administered once a day after breakfast.
  After randomization, the drug for clinical trials is taken once a day (total of 4 tablets) for 8 weeks.
  Other Names: Candesartan 8mg
  Arms: SPC3001
Drug: SPC4001 — Drugs for clinical trials are orally administered once a day after breakfast.
  After randomization, the drug for clinical trials is taken once a day (total of 4 tablets) for 8 weeks.
  Other Names: Amlodipine 5mg
  Arms: SPC4001
Drug: SPC4002 — Drugs for clinical trials are orally administered once a day after breakfast.
  After randomization, the drug for clinical trials is taken once a day (total of 4 tablets) for 8 weeks.
  Other Names: Amlodipine 10mg
  Arms: SPC4002
Drug: Placebo — Drugs for clinical trials are orally administered once a day after breakfast.
  After randomization, the drug for clinical trials is taken once a day (total of 4 tablets) for 8 weeks.

SUMMARY:
This study purpose is to determine the appropriate combination drug dose by comparing safety and efficacy with placebo, candesartan, and amlodipine monotherapy after 8 weeks of administration of SPC1001 to patients with essential hypertension.

DETAILED DESCRIPTION:
This clinical trial is a randomized, double-blind, parallel design, placebo and active drug comparison, and multicenter clinical trial to evaluate the safety and efficacy of investigational drugs after 8 weeks of administration.

Subjects who meet the selection and exclusion criteria should take a placebo for 2 weeks during the run-in period and run a lifestyle improvement program in parallel.

However, if you are already taking antihypertensive drugs at the time of screening, you should stop taking your existing antihypertensive drugs for at least 4 weeks from before the run-in period to the time of randomization to avoid affecting the clinical trial results.

Subjects who meet the final selection and exclusion criteria at the end of the run-in period are randomly assigned 1:1:1:1:1:1:1:1 to each administration group, receive a prescription for clinical trial drugs, and administer for 8 weeks in a double-blind manner.

Encourage the subjects to continuously perform the lifestyle improvement program for 8 weeks during the administration of the clinical investigational drug and visit the testing institution at 4 and 8 weeks during the 8-week trial period, excluding randomized visits, to check the efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women between the ages of 19 and 75
2. Those whose blood pressure measured at the time of screening meets the following criteria 2.1 Not taking antihypertensive drugs (Naïve): 140 mmHg ≤ MSSBP (mean sitting SBP) < 180 mmHg 2.2 If you are taking antihypertensive drugs or have diabetes or chronic kidney disease: 130 mmHg ≤ MSSBP < 180 mmHg
3. Those whose blood pressure measured at the time of randomization meets the following criteria 3.1. 140 mmHg ≤ MSSBP < 180 mmHg 3.2. Or patients with diabetes or chronic kidney disease 130 mmHg ≤ MSSBP < 180 mmHg (However, patients with chronic kidney disease who have clinically significant albuminuria or proteinuria within 6 months)
4. Those who voluntarily agreed to participate in this clinical trial and signed the consent form

Exclusion Criteria:

1. Those whose blood pressure measured at screening and randomization is MSDBP (Mean Sitting DBP) ≥ 110 mmHg
2. Patients who showed a difference of SBP 20 mmHg or more and DBP 10 mmHg or more in blood pressure measured 3 times in both arms at screening
3. Patients with a history of secondary hypertension or any history of suspected secondary hypertension (aortic stenosis, primary hyperaldosteronemia, renal artery stenosis, Cushing's disease, pheochromocytoma, polycystic kidney disease, etc.)
4. Patients with symptomatic orthostatic hypotension
5. Patients requiring concomitant administration of other antihypertensive drugs in addition to investigational drugs during clinical trial participation (Diuretics, β-blockers, ACE inhibitors, Angiotensin II Receptor Blocker, Calcium Channel Blockers, α-blockers, Renin Inhibitors, Vasodilators, etc.)
6. Patients with the following past medical history/comorbidities at the screening visit 6.1. Uncontrolled diabetic patients with HbA1c ≥ 9% 6.2. Patients with severe heart disease (heart failure (NYHA class 3 and 4)), ischemic heart disease (unstable angina, acute myocardial infarction) within 6 months of screening, peripheral vascular disease, percutaneous coronary angioplasty or coronary artery bypass surgery ruler) 6.3. Patients with clinically significant ventricular tachycardia, atrial fibrillation, atrial flutter, or other arrhythmias determined by the investigator to be clinically significant 6.4. Patients with hypertrophic obstructive cardiomyopathy, severe obstructive coronary artery disease, hemodynamically significant aortic stenosis, stenosis on the aortic or mitral valve 6.5. Patients with the severe cerebrovascular disorder (stroke, cerebral infarction, cerebral hemorrhage, etc. within 6 months of screening) 6.6. Patients with known moderate or malignant retinopathy (retinal hemorrhage within 6 months of screening, visual impairment, retinal microaneurysm) 6.7. Patients with wasting disease, autoimmune disease, connective tissue disease 6.8. Patients with gastrointestinal diseases and surgeries that may affect drug absorption, distribution, metabolism, and excretion, current active gastritis, gastrointestinal/rectal bleeding, gastric ulcer, pancreatic dysfunction such as pancreatitis, active inflammatory bowel syndrome within 12 months of screening Back (However, simple appendectomy and hernia surgery are excluded) 6.9. Patients with hereditary angioedema or with a history of angioedema when treated with ACE inhibitors, renin inhibitors, or angiotensin II receptor antagonists 6.10. cholestatic disease patient 6.11. shock patient 6.12. Patients with anuria 6.13. Patients with symptomatic hyperuricemia (history of gout or uric acid stones) 6.14. Patients with a history of malignant tumors including leukemia and lymphoma within 5 years of screening (however, those who have been evaluated as having complete response after treatment and have not relapsed within 2 years of screening, or malignant tumors that have occurred are the only Those with basal cell carcinoma or squamous cell carcinoma of the skin can participate in this test) 6.15. Patients with any chronic inflammatory condition requiring chronic anti-inflammatory treatment
7. Persons whose laboratory test results at the screening visit fall under the following 7.1. Those whose ALT or AST levels are more than 3 times the upper limit of normal organ 7.2. Those whose serum creatinine level is 1.5 times or more of the upper limit of normal organ 7.3. Patients with renal impairment with severe renal failure with Creatinine Clearance (CrCl) < 30 mL/min or eGFR < 30 ml/min/1.73 m2 7.4. Hypokalemia (Serum K < 3.5 mmol/L) 7.5. Persons with hyperkalemia (Serum K > 5.5 mmol/L) 7.6. Those with hyponatremia (Serum Na < 135.0 mmol/L) 7.7. Those with hypercalcemia (Serum Ca > 2.75 mmol/L or 11 mg/dL)
8. Those with genetic problems such as galactose intolerance, Lapp lactase deficiency, or glucose-galactose malabsorption
9. Persons with or suspected of drug or alcohol abuse
10. Pregnant or lactating women
11. Women and men of childbearing potential who do not agree to use a combination of effective or medically acceptable contraceptive methods* for the duration of the clinical trial and 4 weeks after administration of the last investigational drug

    * Taking birth control pills or implanting hormones, implanting intrauterine devices or intrauterine systems, double-blocking methods (both male (condom) and female (contraceptive diaphragm, vaginal sponge or cervical cap) using a contraceptive device), sterilization ( vasectomy, tubal ligation, etc.)
12. Persons with a history of hypersensitivity to clinical investigational drug components and other dihydropyridine drugs, thiazide drugs, or sulfonamide derivatives
13. Those who participated in another clinical trial within 4 weeks before the screening visit and received the investigational drug
14. Others who are judged to be unable to participate in clinical trials cording to the judgment of the investigator

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 253 (Actual)
Dates: Start 2022-03-25 (Actual); Primary Completion 2022-11-27 (Actual); Study Completion 2023-01-27 (Actual)

PRIMARY OUTCOMES:
MSSBP measures the amount of change after 8 weeks from baseline | 8 weeks from baseline
  MSSBP measures the amount of change after 8 weeks from baseline

SECONDARY OUTCOMES:
MSSBP measures the amount of change after 4 weeks from baseline | 4 weeks from baseline
  MSSBP measures the amount of change after 4 weeks from baseline
MSDBP measures the amount of change after 4 weeks, 8 weeks from baseline | 4, 8 weeks from baseline
  MSDBP measures the amount of change after 4 weeks, 8 weeks from baseline
blood pressure normalization rate | 4, 8 weeks from baseline
  The Proportion of subjects who reached target blood pressure at 4 and 8 weeks of administration of the clinical trial drug
blood pressure response rate | 4, 8 weeks from baseline
  The proportion of subjects whose MSSBP decreased by 20 mmHg or more and/or MSDBP decreased by 10 mmHg or more compared to baseline at 4 or 8 weeks after administration of the clinical trial drug

CONTACTS AND LOCATIONS:
Locations (1):
- CHA Gangnam Medical Center, CHA University, Seoul, Gangnam, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shin J, Kim S, Han K, Kim M, Ahn Y, Sohn I, Kim K, Cha D, Hong S, Cho E, Lee H, Pyun W, Youn H, Kim W, Rhee M, Lee J, Ha J, Choi J, Yoo B, Jeong J, Chung W, Jeong Y, Kim C. Multicenter, Randomized, Double-Blind, Parallel, Phase 2 Clinical Trial to Compare and Evaluate the Efficacy and Safety of SPC1001 and Monotherapy in Patients With Essential Hypertension. Clin Ther. 2025 Dec;47(12):1113-1123. doi: 10.1016/j.clinthera.2025.10.001. Epub 2025 Oct 28. PMID 41162308
- See also: From epidemiological transition to modern cardiovascular epidemiology: hypertension in the 21st century — https://www.semanticscholar.org/paper/From-epidemiological-transition-to-modern-in-the-Blacher-L%C3%A9vy/30ae7ff48d49b03b7ba4a4c4533e52d187ab0dc3
- See also: When should antihypertensive drug treatment be initiated and to what levels should systolic blood pressure be lowered? A critical reappraisal — https://journals.lww.com/jhypertension/Abstract/2009/05000/When_should_antihypertensive_drug_treatment_be.3.aspx